CLINICAL TRIAL: NCT05787873
Title: A Clinical Trial to Compare and Evaluate the Safety and Bioequivalence of After Concomitant Administration of "SIPS-2209-2" and "SIPS-2209-3" and Single Administration of "SIPS-2209-1" in Healthy Adult Volunteers in Fasting Conditions.
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetics and Safety of SIPS-2209-1 in Healthy Korean Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samik Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIPS
Record Dates: First submitted 2023-03-05; First posted 2023-03-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: diabetes mellitus; Fixed-dose combination; Bioequivalence
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A (Experimental): Period 1: SIPS-2209-1 - A single oral dose of 1 tablet under fasting condition
  Period 2: SIPS-2209-2, SIPS-2209-3 - A single oral dose of 2 tablets under fasting condition
  Interventions: Drug: SIPS-2209-1; Drug: SIPS-2209-2, SIPS-2209-3
- Sequence B (Experimental): Period 1: SIPS-2209-2, SIPS-2209-3 - A single oral dose of 2 tablets under fasting condition
  Period 2: SIPS-2209-1 - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: SIPS-2209-1; Drug: SIPS-2209-2, SIPS-2209-3

INTERVENTIONS:
Drug: SIPS-2209-1 — QD, PO
Drug: SIPS-2209-2, SIPS-2209-3 — QD, PO

SUMMARY:
The goal of this clinical trial is to evaluate of bioequivalence between fixed-dose combination and co-administration of the individual components under fasting conditions in healthy Korean volunteers.

DETAILED DESCRIPTION:
40 healthy subjects are administered the corresponding drug for each period, and the drug wash-out period is set to 7 days. Pharmacokinetic samples are collected for up to 36 hours. Pharmacokinetic parameters are compared to evaluate bioequivalence, and additionally, safety are evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Male for body weight ≥50 kg, female for body weight ≥45 kg
3. Calculated body mass index (BMI) of 18 to 30 kg/m2
4. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
5. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serology, urology) and ECG results at screening.
6. Those who agree to contraception during the participation of clinical trial.
7. Those who agrees to exclude the possibility of pregnancy by using a medically accepted method of contraception from the first administration of investigational medicine to 7 days after the last administration of investigational medicine

Exclusion Criteria:

1. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
2. Those who take barbiturate and any related drugs which may cause induction or inhibition of drug metabolism within 1 month and those who take drug could affect to clinical trial within 10 days before the first administration of investigational products.
3. Those who donated whole blood or apheresis within 8 weeks or 2 weeks respectfully, or received blood transfusion within a month.
4. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
5. Those who exceed an alcohol and cigarette consumption criteria write below within 1 month before the first administration of investigational products.

   * Alcohol: Man - 21 glasses/week, Woman - 14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL)
6. Patients with the following diseases

   * Patients with known hypersensitivity reactions such as anaphylaxis or angioedema to investigational drugs and components
   * Patients with pancreatitis
   * Patients with heart failure or a history of heart failure
   * Patients with active bladder cancer or a history of bladder cancer
   * Patients with hepatic impairment
   * Patients with severe renal impairment
   * Patients with diabetic ketoacidosis, diabetic coma and pre-coma, patients with type 1 diabetes
   * Before and after surgery, patients with severe infections, patients with severe trauma
   * Patients with gross hematuria not investigated
   * Patients with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
7. Those who are deemed insufficient to participate in this clinical trial by investigators.
8. Woman who are pregnant or breastfeeding.
9. Those who have a history of clinically significant mental illness

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
AUCt of SIPS-2209-1 | predose (0 hours), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 hours
  AUCt: Area under the concentration-time curve from time zero to time
Cmax of SIPS-2209-1 | predose (0 hours), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 hours
  Cmax: Maximum plasma concentration of the drug

SECONDARY OUTCOMES:
AUCinf of SIPS-2209-1 | predose (0 hours), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 hours
  AUCinf : AUC from time 0 to infinity
CL/F of SIPS-2209-1 | predose (0 hours), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 hours
  CL/F : Clearance
Tmax of SIPS-2209-1 | predose (0 hours), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 hours
  Tmax : Time to maximum plasma concentration of drug
t1/2 of SIPS-2209-1 | predose (0 hours), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 hours
  t1/2 : Terminal half-life
Vd/F of SIPS-2209-1 | predose (0 hours), 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36 hours
  Vd/F : Volume of distribution based on the terminal phase

CONTACTS AND LOCATIONS:
Overall Officials: Young Ee KWON, Ph.D, Study Director — Samik Pharmaceutical Co. Ltd.
Locations (1):
- Samik Pharmaceutical Co. Ltd., Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No